CLINICAL TRIAL: NCT05119036
Title: Adjuvant Treatment Deintensification After Transoral Surgery for Human Papillomavirus-Positive Squamous Cell Carcinoma of the Oropharynx
Brief Title: Adjuvant Treatment Deintensification After Transoral Surgery for Human Papillomavirus-Positive Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael W. Sim, Assistant Professor of Otolaryngology, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OTHN-CC-IUSCCC-0756
Record Dates: First submitted 2021-09-22; First posted 2021-11-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: transoral surgery; HPV
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Observation (No Intervention): If patients have negative margins and have all negative nodes or only a single positive node, patients will be placed in the observation arm and will not receive further adjuvant treatment, only postoperative follow-up visits and a surveillance visit 3 months after surgery with a CT or PET-CT.
- Adjuvant Radiation 44 Gray (Experimental): If patients have 4 or fewer positive nodes and 2 mm or less of cancer spread extending outside the lymph nodes, patients will receive 44 gray fractions (the full dose of radiation divided into smaller doses) of adjuvant radiation.
  Interventions: Radiation: 44 doses of radiation
- Adjuvant Radiation 54 Gray (Experimental): If patients have 4 or fewer positive nodes with greater than 2 mm of cancer spread extending outside the lymph nodes or 5 or more positive nodes with 2 mm or less of cancer spread extending outside the lymph nodes, patients will receive 54 gray fractions (the full dose of radiation divided into smaller doses) of adjuvant radiation.
  Interventions: Radiation: 54 doses of radiation

INTERVENTIONS:
Radiation: 44 doses of radiation — Patients will receive 44 gray in 22 fractions to the operative bed, including the primary tumor site and dissected nodal basin. Patients will receive 40 gray in 22 fractions to undissected areas of the neck at low-risk for occult disease.
  Arms: Adjuvant Radiation 44 Gray
Radiation: 54 doses of radiation — Patients will receive 54 gray in 27 fractions to the operative bed, including the primary tumor site and dissected nodal basin. Patients will receive 50 gray in 27 fractions to undissected areas of the neck at low-risk for occult disease.
  Arms: Adjuvant Radiation 54 Gray

SUMMARY:
Oropharyngeal squamous cell carcinoma (OPSCC), commonly known as throat cancer or tonsil cancer, has seen a dramatic rise in incidence over the last twenty years. There are two types of OPSCC: human papillomavirus-positive (HPV+) and human papillomavirus-negative (HPV-). People with OPSCC, regardless of their type, typically receive standard treatment with a combination of chemotherapy, radiation therapy, and surgery. Due to the intensity of standard treatment, survivors may experience unwanted long-term side effects. The goal of this research study is to see if intensifying (stopping or scaling back) treatment still provides the same, or perhaps even better, results when compared to standard treatment.

DETAILED DESCRIPTION:
Oropharyngeal squamous cell carcinoma (OPSCC) has seen a dramatic rise in incidence over the last two decades. This is largely due to the increased incidence of human papillomavirus-positive (HPV+) malignancy within the oropharynx. In fact, HPV-positive (HPV+) OPSCC has surpassed cervical cancer as the most common HPV related malignancy in the United States. Thus, with the current widespread prevalence of HPV infection, OPSCC will continue to be a major factor in cancer treatment in the national healthcare landscape for years to come.

Fortunately, patients with HPV+ OPSCC have substantially improved treatment response and overall survival (OS) compared to those with HPV-negative malignancy. Prior surgical procedures to remove tumors within the oropharynx were very invasive and highly morbid, requiring face and neck incisions along with mandibulotomy and pharyngotomy approaches. Therefore, treatment paradigms shifted to favor concurrent chemoradiation as the primary treatment modality over primary surgery. However, the acute and long-term toxicity of chemoradiation can be significant, including swallow dysfunction, speech disturbance, taste disturbance, mucositis, xerostomia, fibrosis, osteoradionecrosis, neutropenia, neurotoxicity, and dental disease. With improved survival rates associated with HPV+ OPSCC, more patients are surviving their disease and experiencing these side effects, negatively impacting quality of life (QOL).

With early studies establishing the more favorable prognosis associated with HPV+ OPSCC9, the staging system for OPSCC was completely changed, with HPV+ OPSCC given its own separate system from its HPV negative counterpart. Even with higher nodal burden, HPV+ OPSCC has lower stages, reflecting improved treatment response of this disease. Notably, this reclassification omitted extranodal extension (ENE) as a component of the N staging.

The advent of transoral robotic surgery (TORS) via the da Vinci Surgical System, and other minimally invasive techniques, has reaffirmed surgical therapy as a primary treatment option, as these approaches provide quicker recovery times and confer less morbidity to patients. The safety and oncologic efficacy of TORS has been well-established for the treatment of OPSCC. For example, in one large multi-institutional study of 410 patients undergoing TORS, the 2-year locoregional control rate was 91.8%, disease-specific survival rate 94.5%, and overall survival 91%13. Now, the majority of patients undergo surgery for T1-T2 disease (82%) in the United States according to an analysis of the National Cancer Data Base.

The goal of primary surgical therapy is to minimize long term toxicity by eliminating the need for chemotherapy, decreasing radiation intensity to adjuvant doses, and in some cases, obviating the need for adjuvant therapy altogether while still providing equivalent or even superior oncologic results compared to standard chemoradiation. The resulting effects are improvement in functional outcomes and QOL for patients surviving their disease. The prevailing treatment philosophy within head and neck oncology is that further deintensifying treatment could still provide equivalent oncologic outcomes, while further lowering toxicity profiles and improving functional outcomes even more. There are now numerous trials investigating deintensification in an attempt to minimize the morbidity incurred by patients, and strategies have varied greatly. But still, there is no level I evidence for deintensification, and certainly, no consensus on the best strategies for treatment moving forward in the near future.

One such trial focusing on surgical therapy with de-escalated radiotherapy is ECOG-3311, a randomized phase II trial which focuses on a primary surgical approach for cT1-2 N1-2b (as per AJCC 7th edition) HPV+ OPSCC. The study de-escalates the adjuvant radiation dose to 50 gray for intermediate risk patients based on surgical pathology results. But even in this study, nearly a third of the patients received adjuvant chemoradiation therapy which raises concerns for even worse functional outcomes in those patients receiving triple modality therapy (surgery, radiation, and chemotherapy). The final results of this study are still pending.

In another phase II trial, the Mayo Clinic group randomized patients to either standard adjuvant treatment or deintensified treatment after TORS, administering between 30 to 36 Gray of radiation along with concurrent docetaxel infusion in the latter group. In that study, the most important risk factors for progression were higher T stage, pN2 disease (5 or more positive nodes), and the presence of ENE. Moreover, those with pN2 and ENE were at high risk for distant failure. The 3-year progression-free survival (PFS) rate for the deintensified cohort was 87%, compared to the standard cohort PFS of 90%. The group still concluded that even patients with high risk features could still benefit from deintensification as both groups did poorly from a distant disease standpoint.

Other studies have shown the significance of having pN2 disease, as well, with associated higher risk for distant disease. In a large multi-institutional study, patients with HPV+ OPSCC who underwent primary surgical therapy and found to have 4 or fewer positive nodes had improved 5-year overall survival compared to those with 5 or more positive nodes (89% vs 71%, respectively). This was the basis for the change in staging for the AJCC 8th edition in which pN1 was designated for 1 to 4 positive nodes and pN2 for 5 or more positive nodes. Moreover, ENE was removed as a stratifying factor in the N staging for HPV+ OPSCC, as previously mentioned. The significance of ENE remains a point of contention, and there is currently no level I evidence for the optimal management of ENE in the adjuvant setting for surgically managed HPV+ OPSCC. Often times, chemotherapy is recommended if ENE is identified, but the addition of the third modality significantly worsens toxicity profile without assuredly providing benefit. Recent NCCN guidelines recommend adjuvant radiation of 44 to 50 gray in low risk, 54 to 63 gray in intermediate risk, and 60 to 66 gray for high risk patients, with or without the addition of chemotherapy.

There is no doubt about the clinical impact of HPV+ OPSCC in the future of the national healthcare system. Despite this, there is still no consensus on the best treatment strategies for this disease. The investigators at IU have performed over 125 TORS operations in the last four years since the inception of the Robotic Head and Neck Surgery Program with excellent oncologic outcomes. The investigators anticipate the surgical volume to continue to grow as the treatment paradigm shifts back to primary surgery and the incidence of HPV+ OPSCC continues to rise. Thus, the purpose of this phase II prospective trial is to assess the safety and efficacy of deintensification after surgical therapy in early stage HPV+ OPSCC by evaluating oncologic outcomes, toxicity profiles, functional outcomes, and QOL measures, and compare these factors to historical controls. This protocol also seeks to more clearly define the setting and safety of eliminating of chemotherapy in the adjuvant setting after transoral surgery for HPV+ OPSCC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years old at the time of informed consent.
* Ability to provide written informed consent and HIPAA authorization.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (refer to Appendix).
* Primary tumor of the oropharynx (palatine tonsil, tongue base, soft palate, lateral or posterior walls of oropharynx).
* Histopathologically confirmed squamous cell carcinoma.
* HPV+ tumor, as determined by p16, in-situ hybridization, or real-time polymerase chain reaction.

  * Note: If patients present who have unconfirmed p16/HPV positive disease but have clinical findings that indicate a high probability of HPV positive disease, these patients can be deemed eligible after testing is performed at post-surgery.
* Resectable and accessible tumor with high probability of achieving negative margins.
* Smokers and non-smokers included.
* Tumor stage (AJCC 8th edition): T1 or T2.
* Nodal stage (AJCC 8th edition): N0, N1 or N2.
* Mobile neck nodes on physical exam if N positive.
* Subjects with synchronous primaries included.
* Subjects with unknown primaries included if primary is definitively identified and resectable with negative margins or if the palatine and lingual tonsils are thoroughly resected and pathologically proven to be negative for a primary.

Exclusion Criteria:

* Serious medical condition preventing general anesthesia for surgery.
* Inability to complete full course of radiation treatment or attend follow-up visits.
* History of previous head and neck radiation or previous head and neck cancer within 3 years.
* Distant metastatic disease present.
* Prior invasive malignant disease within 3 years, with the exception of non-melanoma skin cancer and thyroid cancer, unless patient is deemed cured or disease free, in which case patient may be included in the study.
* Lactating or pregnant women. Women of childbearing potential must have a negative pregnancy test within 60 days of protocol registration. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless the patients meet one of the following criteria:

  1. Has undergone a hysterectomy or bilateral oophorectomy; or
  2. Has been naturally amenorrheic for at least 24 consecutive months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | Day 1 until death, assessed up to 2 years
  Time from surgery to first disease recurrence or death from any cause

SECONDARY OUTCOMES:
Loco-regional control | Day 1 - Day 365
  Rate of subjects with no recurrence at primary oropharyngeal site or in the neck nodal basins within 1 year
Overall survival | Day 1 until death, assessed up to 2 years
  Time of surgery until death from any cause
Distant metastasis rates | Day 1 - Day 365
  Assessed by tissue diagnosis or radiographically of recurrent disease at sites away from the primary tumor and neck nodal basins within 1 year
Toxicity from radiation | Day 1 - Day 180
  Toxicity within 6 month as assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) version 5.0
Swallowing-related Quality of Life | at 3 months, 6 months, 1 year, and 2 year post-treatment
  Assessed using MDADI
Gastrostomy tube dependence rates | Day 365
  Assessed by confirmation of feeding tube in-situ in subject and being utilized for nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sim, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No